CLINICAL TRIAL: NCT01174485
Title: Effects of Liposuction and Exercise Training on Metabolism, Lipid Profile and Adiposity in Women
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Fabiana Braga Benatti, Escola de Educação Física e Esporte da Universidade de São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EEFEUSP-LIPO
Record Dates: First submitted 2010-06-25; First posted 2010-08-03 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-04

CONDITIONS: Healthy Subjects
Keywords: Liposuction; exercise; metabolism; adiposity
MeSH Terms: conditions — Motor Activity; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise (Experimental): exercise plus liposuction
  Interventions: Procedure: exercise
- sedentary (No Intervention): physical inactivity plus liposuction

INTERVENTIONS:
Procedure: exercise — combined resistance and aerobic training
  Arms: exercise

SUMMARY:
Liposuction is the most popular aesthetic surgery in Brasil and worldwide. Evidence showing that adipose tissue is a metabolically active tissue led to the suggestion that liposuction could be a viable method for the improvement of metabolic profile through the immediate loss of adipose tissue. Studies about the effects of liposuction on metabolic profile are conflicting. A few studies report the improvement of insulin sensitivity, inflammatory markers and lipid profile, others observe no changes and a few report the worsening of metabolic profile. In addition, animal studies show a compensatory growth of intact adipose tissue in response to lipectomy. Physical exercise improves insulin sensitivity, lipid profile, inflammatory balance, adipose tissue distribution and increases or preserves free fat mass. Therefore, liposuction and physical exercise seem to act on similar tissues of the body. To the investigators knowledge, there are no studies about the associated effects of liposuction and exercise in humans. However, one can suggest that exercise training associated with liposuction could: [1] attenuate or block the possible fat recovery or compensatory growth; [2] block or reverse the possible harmful effects of liposuction; or [3] exert an additive or synergistic effect to the possible beneficial effects induced by liposuction on metabolic and hormonal profile and inflammatory balance.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 35-year old healthy subjects with a BMI of 22 to 28 Kg/m2;
* Non-smokers;
* Present stable body weight for 6 months (without variations exceeding 4 kg);
* Be in use contraceptive pill for at least 6 months;

Exclusion Criteria:

* Health problems that impede surgery or exercise training;
* Be in chronic use of antibiotics or antiinflammatory medication.

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Body composition | 2 months post-intervention
  Body composition will be assessed by hydrostatic weighing in order to measure fat and lean mass and by computer tomography, in order to measure abdominal total, subcutaneous and visceral fat areas and femoral and pelvic subcutaneous fat areas.
Body composition | 6 months post-intervention
  Body composition will be assessed by hydrostatic weighing in order to measure fat and lean mass and by computer tomography, in order to measure abdominal total, subcutaneous and visceral fat areas and femoral and pelvic subcutaneous fat areas.

SECONDARY OUTCOMES:
Insulin Sensitivity | 2 months post-intervention
  Insulin sensitivity will be assessed by an oral glucose tolerance test
Total cholesterol, LDL-c, HDL-c, VLDL-c and triacylglycerol plasma levels | 2 months post-intervention
Cytokine plasma levels - IL-6, TNF-alpha, IL-10, leptin and adiponectin levels | 2 months post-intervention
Insulin Sensitivity | 6 months post-intervention
  Insulin sensitivity will be assessed by an oral glucose tolerance test
Total cholesterol, LDL-c, HDL-c, VLDL-c and triacylglycerol plasma levels | 6 months post-intervention
Cytokine plasma levels - IL-6, TNF-alpha, IL-10, leptin and adiponectin levels | 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Antonio H Lancha Jr, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Escola de Educação Física e Esporte da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Benatti F, Solis M, Artioli G, Montag E, Painelli V, Saito F, Baptista L, Costa LA, Neves R, Seelaender M, Ferriolli E, Pfrimer K, Lima F, Roschel H, Gualano B, Lancha A Jr. Liposuction induces a compensatory increase of visceral fat which is effectively counteracted by physical activity: a randomized trial. J Clin Endocrinol Metab. 2012 Jul;97(7):2388-95. doi: 10.1210/jc.2012-1012. Epub 2012 Apr 26. PMID 22539589